CLINICAL TRIAL: NCT06004193
Title: Holiday Season Weight Change During Islamic Holidays and Effect of Exercise on Body Weight and Body Composition
Brief Title: Holiday Season Weight Change During Islamic Holidays
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Goktas, Principal Investigator, Hacettepe University
Other Study IDs: GO 16/307
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Body Weight Changes
Keywords: Holiday weight gain; Fasting; Body composition
MeSH Terms: conditions — Body Weight Changes; Fasting | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular Exercisers: The group of regular exercisers includes individuals who engage in at least 150 minutes of exercise per week according to World Health Organization criteria.
  Interventions: Behavioral: Exercise
- Non-exercisers: The group of non-exercisers includes individuals who do not have a habit of engaging in regular exercise.

INTERVENTIONS:
Behavioral: Exercise — At least 150 minutes of exercise in a week
  Groups: Regular Exercisers

SUMMARY:
The study involved 30 regular exercisers and 33 non-exercisers. Food records were collected five times: before the holiday season, before Ramadan, during Ramadan, during Ramadan Feast, and after Ramadan Feast, including the Eid al-Adha period. Anthropometric measurements were taken before and after holidays: initially before Ramadan and again after Eid al-Adha. Physical activity was recorded for both groups: once before Ramadan for non-exercisers and twice (on exercise and rest days) for exercisers.

DETAILED DESCRIPTION:
The purpose of this study is to determine the changes in nutrient consumption during the holiday season and to assess the changes in body weight, body composition, and blood pressure of exercising and non-exercising individuals at the end of this season. In the United States of America, the holiday season is the period between Thanksgiving and New Year's Day. In Turkey, the holiday season is defined as the period between the Feast of Ramadan and the Feast of Sacrifice. A total of 30 individuals who regularly exercise and 33 who do not exercise participated in the study. In this study, 3-day food consumption records were taken from the participants five times; before the holiday season, before Ramadan, during Ramadan, during Ramadan Feast, after Ramadan Feast, and during the Eid al-Adha period. The anthropometric measurements of the participants were measured before and after the holidays. The first measurement was taken before Ramadan, and the second was taken after Eid al-Adha. Physical activity was recorded in the pre-Ramadan period, once for non-exercising participants, and twice for exercising participants, on exercise and rest days.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 45 years
* Body mass index (BMI) between 18.5-40.0kg/m2
* Observing the Islamic holiday season.

Exclusion Criteria:

* Pregnant or lactating women
* Chronic metabolic diseases including type 1 or type 2 diabetes, any type of cancer, cardiovascular diseases
* 5kg of weight gain or loss in the last 3 months
* Planning to lose weight or following a specific diet
* Exercising >300min/week
* Medication use that might affect body weight or composition

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants were recruited from a local activity center, which includes a gym as well as art studios, via bulletin board announcement.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Body weight | 4 months
  Body weight measurements
Body fat percentage | 4 months
  Body fat percentage measured with bioelectrical impedance analysis
Dietary intake | 4 months
  24-hour dietary recall questionnaires were administered by researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goktas, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Nutrition and Dietetics Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No